CLINICAL TRIAL: NCT01782001
Title: Evaluation of the Impact of Vitamin A and Zinc Supplementation on Malarial Morbidity in Ghana
Brief Title: Evaluation of Vitamin A and Zinc Supplementation on Malarial Morbidity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kintampo Health Research Centre, Ghana (Other)
Collaborators: International Atomic Energy Agency (Other Government); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AMANI
Record Dates: First submitted 2013-01-27; First posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Malaria; Malnutrition
Keywords: Vitamin A; Zinc; Malaria; Morbidity; MRDR
MeSH Terms: conditions — Malaria; Malnutrition | interventions — Vitamin A; Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin A and zinc (Experimental): combination of vitamin A and zinc supplements
  Interventions: Dietary Supplement: vitamin A and zinc
- Vitamin A and placebo (Active Comparator): vitamin A with placebo
  Interventions: Dietary Supplement: vitamin A

INTERVENTIONS:
Dietary Supplement: vitamin A — vitamin A with placebo
  Arms: Vitamin A and placebo
Dietary Supplement: vitamin A and zinc — combination of vitamin A and zinc supplements
  Arms: Vitamin A and zinc

SUMMARY:
The purpose of this study was to determine whether young children receiving Vitamin A and Zinc supplements will have a lower incidence of symptomatic malaria than similar children receiving vitamin A supplements alone.

DETAILED DESCRIPTION:
The aim of our study was to determine the impact of the combination of vitamin A and zinc supplements on malaria morbidity in young children. The primary objective was to determine the effect of vitamin A alone vs. vitamin A and zinc supplements on the incidence of clinical malaria. The specific objectives were to determine the effect of vitamin A alone vs. vitamin A and zinc supplements on changes in anthropometric measurements specifically weight and length/height and to assess the effect of the study interventions on the incidence of anemia, diarrhea and pneumonia. It also assessed the tolerability of the supplements and determined the change in zinc status by measuring plasma zinc concentration using atomic absorption spectrometry before and at the end of the intervention. The study also determined the change in vitamin A status as assessed by the modified relative dose response (MRDR) test during and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 - 24 months
* Child's guardian is willing to provide informed consent
* Child's family plans to remain resident in the study areas during the study period

Exclusion Criteria:

* Clinical evidence of vitamin A deficiency
* Severe acute malnutrition
* Severe illness
* Child aged <6 months or >24 months
* Receipt of vitamin A supplement within the last three months

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
incidence of clinical malaria attacks | 6 months

SECONDARY OUTCOMES:
changes in weight and height/length | baseline and 6 months
  Enrollment and end of supplementation
changes in vitamin A and zinc nutritional status within and between the groups | baseline and 6 months
  enrollment and end of supplementation
change in prevalence of anemia | baseline and 6 months
  enrollment and end of supplementation
the incidence of diarrhea and pneumonia | 1 time per week up to 6 months
  1 time/week, enrollment to end, total:24

CONTACTS AND LOCATIONS:
Overall Officials: Seth Owusu-Agyei, PhD, Principal Investigator — Kintampo Health Research Centre, Ghana
Locations (1):
- Kintampo Health Research Centre, Kintampo, Brong Ahafo, Ghana